CLINICAL TRIAL: NCT01627379
Title: An Open-label, Randomized Phase III Trial of Cisplatin and 5-fluorouracil With or Without Panitumumab for Patients With Nonresectable, Advanced or Metastatic Esophageal Squamous Cell Cancer
Brief Title: Cisplatin and 5-FU +/- Panitumumab for Patients With Nonresectable,Advanced or Metastatic Esophageal Squamous Cell Cancer
Acronym: POWER
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision due to recommendation of the IDMC.
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Amgen (Industry); Assign Data Management and Biostatistics GmbH (Other); Assign Clinical Research GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POWER / AIO-STO-0309; 2010-020606-15 (EudraCT Number)
Record Dates: First submitted 2012-06-13; First posted 2012-06-25 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Esophageal Squamous Cell Cancer
Keywords: nonresectable; advanced; metastatic esophageal squamous cell cancer; Panitumumab
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Cisplatin; Fluorouracil; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Cisplatin, 5-Fluorouracil (Active Comparator): Chemotherapy will be administered every 3 weeks until progression of disease or any other reason for treatment withdrawal is fulfilled.
  Interventions: Drug: Cisplatin, 5-FU
- Arm B: Cisplatin, 5-Fluorouracil and Panitumumab (Experimental): Chemotherapy plus Panitumumab will be administered every 3 weeks until progression of disease or any other reason for treatment withdrawal is fulfilled.
  Interventions: Drug: Panitumumab

INTERVENTIONS:
Drug: Cisplatin, 5-FU — Arm A: Cisplatin 80 mg/m2 IV infusion over 2 hours on Day 1, followed by 5-FU 1000 mg/m2 IV daily as continuous infusion over 24 hours, Day 1-4.
  Chemotherapy will be administered every 3 weeks until progression of disease or any other reason for treatment withdrawal is fulfilled.
  Arms: Arm A: Cisplatin, 5-Fluorouracil
Drug: Panitumumab — Arm B: Cisplatin 80 mg/m2 IV infusion over 2 hours on Day 1, followed by 5-FU 1000 mg/m2 IV daily as continuous infusion over 24 hours, Day 1-4.
  Panitumumab will be administered on Day 1 of each treatment cycle at a dose of 9 mg/kg prior to administration of chemotherapy.
  Each treatment cycle is defined as 21 days. Patients are treated until progression of disease occurs or any other reason for treatment withdrawal is fulfilled.
  Arms: Arm B: Cisplatin, 5-Fluorouracil and Panitumumab

SUMMARY:
More than 50% of patients with esophageal cancer have locally advanced or metastatic disease at presentation. The use of chemotherapy for this patient group is increasing with the intention of local and distant tumor control, improving quality of life and prolongation of survival.

Previous data suggested not only that EGFR antibody targeted therapy may be safely combined with cisplatin and 5-FU but also may increase the efficacy of standard cisplatin / 5-FU regime.

In the present study, patients with nonresectable, advanced or metastatic esophageal squamous cell cancer (ESCC) will receive chemotherapy or chemotherapy plus panitumumab every 3 weeks until disease progression occurs.

The primary objective is to demonstrate superiority of 5-FU, Cisplatin and Panitumumab over 5-FU and Cisplatin alone in terms of overall survival in esophageal cancer.

DETAILED DESCRIPTION:
More than 50% of patients with esophageal cancer have locally advanced or metastatic disease at presentation. The use of chemotherapy for this patient group is increasing with the intention of local and distant tumor control, improving quality of life and prolongation of survival. The most frequently used agents are 5-fluorouracil, cisplatin, with or without various anthracyclines. Cisplatin plus continuous 5-fluorouracil are the standard of care regimens. Taxanes and anthracyclins are eligible agents for possible future studies, however with higher incidences of toxicities and life threatening complications. Response rates for single agents range from 15%-30%. Combination regimens usually tend to produce higher response rates and occasionally patients achieve complete responses (0%-11%). However, with the combination regimens, the median survival time remains clearly less than 10 months, mostly between 4-8 months [Homs MY et al]. In comparison of different chemotherapy protocols, there was no consistent benefit of any specific chemotherapy regimen. So far, cisplatin combined with 5-fluorouracil is one of the approved standard regimens in esophageal cancer world wide[Medical Research Council Oesophageal Cancer Group]. This so called three-weekly MRC regimen has a better toxicity profile than the four weekly CF regimen given in Central Europe with the higher Cisplatin dose[Lorenzen S et al], but less overall chemotherapy given per 4 months.

Advances in molecular biology and new molecular technologies can possibly contribute to improvement of response to neoadjuvant or palliative therapy in ESCC patients as well. EGFR1 blockade with platinum-based chemotherapy already significantly improved response rates as well as the progression-free and overall survival compared to chemotherapy alone in patients with head and neck tumors, which are also squamous cancers[Vermorken JB et al].

Even more, the Arbeitsgemeinschaft Internistische Onkologie (AIO) has performed a randomized phase II study of the EGFR antibody cetuximab plus cisplatin/5-fluorouracil versus cisplatin/5-fluorouracil alone in first-line metastatic ESCC[Lorenzen S et al]. For a maximum of six 28-day cycles, patients received cisplatin 100 mg/m(2), day 1, plus 5-FU 1000 mg/m(2) days 1-5 (CF), either alone or in combination with cetuximab (CET-CF). The primary endpoint was tumor response. From 62 eligible patients included, 32 receiving CET-CF and 30 CF. Cetuximab weekly did not exacerbate grade 3/4 toxicity, except for rash (6% vs 0%) and diarrhea (16% vs 0%). The overall response rate according to RECIST criteria were 19% and 13% and the disease control rates, were 75% and 57% for the CET-CF and CF arms, respectively. With a median follow-up of 21.5 months, the median progression-free survival was 5.9 and 3.6 months and median overall survival 9.5 and 5.5 months for CET-CF and CF, respectively. No KRAS codon 12/13 tumor mutations were identified in the 37 evaluated samples.

Thus, with respect to the AIO data and in concordance with the head and neck data by Vermorken, EGFR antibody targeted therapy may not only be safely combined with CF, but may also very likely increase the efficacy of standard CF, particularly with regard to a chosen primary endpoint of overall survival. Therefore, the aim of this study is to investigate if the overall survival of patients with squamous cell carcinoma of the esophagus can be prolonged if panitumumab is added to the standard CF chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Male or female ≥18 years of age
3. Histologically proven squamous cell carcinoma of the esophagus, which is not curatively resectable* or locally recurrent disease and both not eligible** for definitive radiochemotherapy, or clearly metastatic disease (Tx, Nx, M1, locally unresectable T4, Nx, M0 or TX, N3, M0)* or residual (post-resection) disease not eligible** for definitive radiochemotherapy

   * resectability has to be defined prior to randomization according to local standards:

   The tumor is considered unresectable due to:

   T-stage, N-stage, performance status/nutritional status, co-morbidity (pulmonary function, other), tumor location upper third of the esophagus, relation to other organs/structures), patient refusal, other reasons.
   * eligibility to definitive radiochemotherapy will be determined according to local standards based on the extent of disease, performance status/nutritional status, co-morbidity (pulmonary function, other), volume of neighboring organs within the radiation field, patient refusal, other reasons.
4. Measurable or non-measurable disease according to RECIST 1.1
5. ECOG 0-1
6. Women of child-bearing potential must have a negative pregnancy test
7. Laboratory requirements

   * Hematology:

     * Absolute neutrophil count ≥1.5x10^9/L
     * Platelet count ≥100x10^9/L
     * Leukocyte count ≥ 3.0x10^9/L
     * Hemoglobin ≥ 9 g/dL or 5.59 mmol/l
   * Hepatic Function:

     * Total bilirubin ≤ 1.5 time the upper normal limit (UNL)
     * AST ≤ 2.5xUNL in absence of liver metastases, or ≤5xUNL in presence of liver metastases
     * ALT ≤ 2.5xUNL in absence of liver metastases, or ≤5xUNL in presence of liver metastases
   * Renal Function:

     * Creatinine clearance ≥ 50 mL/min according to Cockroft-Gault formula
   * Metabolic Function

     * Magnesium ≥ 0.5 mmol/L or 1.2 mg/dL
     * Calcium ≥ 2 mmol/L or 8.0 mg/dL

Exclusion Criteria:

1. Previous chemotherapy of esophageal cancer in the metastatic setting. Previous neoadjuvant chemotherapy or definitive radiochemotherapy with a maximum cumulative dose of 120 mg cisplatin and without recurrence of disease within 4 months after the end of treatment is allowed.
2. Concurrent radiotherapy involving target lesions used for this study. Concurrent palliative radiation for non-target lesions is allowed if other lesions are available outside the involved field. Previous pre- operative or post-operative radiotherapy is allowed.
3. Previous exposure to EGFR-targeted therapy
4. Other previous malignancy with exception of a history of a previous curatively treated basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix or other curatively treated malignant disease without recurrence after at least 5 years of follow-up
5. Known brain metastases unless adequately treated (surgery or radiotherapy) with no evidence of progression and neurologically stable off anticonvulsants and steroids
6. Serious concomitant disease or medical condition that in the judgment of the investigator renders the subject at high risk of treatment complication or reduces the probability of assessing clinical effect.
7. Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year before enrollment
8. Inadequate pulmonary function according to the investigator's judgment, history of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan.
9. Hearing loss ≥ NCI-CTC V.4.03 Grade 3
10. Subject pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment.
11. Subject (male or female) is not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment.
12. Contraindications to receive any platin, 5-FU or panitumumab
13. Concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational drug within 30 days prior to treatment start
14. Known drug abuse/alcohol abuse
15. Peripheral polyneuropathy ≥ NCI-CTC V 4.03 Grade 2
16. Chronic inflammatory bowels diseases
17. Social situations limiting the compliance with the study requirements.
18. History of HIV infection or chonic hepatitis B or C
19. Concurrent treatment with brivudin or sorivudin or its chemically related analogues. There must be at least a 4-week wash-out period between end of treatment with brivudin, sorivudin or its chemically related analogues and start of therapy with 5-FU.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 3 years
  Kaplan-Meier estimate of the median time between date of randomization and the date of death from any cause or the date of last follow-up in case of no documentation of death.
  Comparison of Overall survival of treatment arms "Panitumumab + Chemotherapy" and "Chemotherapy only" in patients with nonresectable, advanced or metastatic ESCC.

SECONDARY OUTCOMES:
Progression-free survival | every 9 weeks from Cycle 1 up to 3 years
  Kaplan-Meier estimate of the median time span between the date of randomization and the date of progression or death due to any cause.
  The difference in progression-free survival between the two treatment arms will be tested.
  Tumor assessments will be performed every 9 weeks during the treatment period.
1-year survival | 1 year
  The difference in 1-year survival between the two treatment arms is determined.
Response rate | every 9 weeks from Cycle 1 up to 3 years
  Best objective response is defined as the best response documented during study. To compare objective response rate between the two treatment arms.
  Tumor Assessments will be performed every 9 weeks during the treatment period.
Overall incidence of patients with adverse events | up to 3 years
  Throughout the treatment period until the End of treatment visit, patients will be assessed for all adverse events. CTCAE V 4.03 will be used for grading.
Quality of life | every 3 weeks for up to 3 years
  EORTC QLQ-C30 questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Markus Möhler, PD Dr., Principal Investigator — I. Medizinische KLinik und Poliklinik, Johannes-Gutenberg-Universität Mainz
Locations (1):
- Johannes-Gutenberg-Universität Mainz, I. Medizinische Klinik und Poliklinik, Mainz, Rhineland-Palatinate, Germany

REFERENCES:
- [Background] Vermorken JB, Mesia R, Rivera F, Remenar E, Kawecki A, Rottey S, Erfan J, Zabolotnyy D, Kienzer HR, Cupissol D, Peyrade F, Benasso M, Vynnychenko I, De Raucourt D, Bokemeyer C, Schueler A, Amellal N, Hitt R. Platinum-based chemotherapy plus cetuximab in head and neck cancer. N Engl J Med. 2008 Sep 11;359(11):1116-27. doi: 10.1056/NEJMoa0802656. PMID 18784101
- [Background] Lorenzen S, Schuster T, Porschen R, Al-Batran SE, Hofheinz R, Thuss-Patience P, Moehler M, Grabowski P, Arnold D, Greten T, Muller L, Rothling N, Peschel C, Langer R, Lordick F. Cetuximab plus cisplatin-5-fluorouracil versus cisplatin-5-fluorouracil alone in first-line metastatic squamous cell carcinoma of the esophagus: a randomized phase II study of the Arbeitsgemeinschaft Internistische Onkologie. Ann Oncol. 2009 Oct;20(10):1667-73. doi: 10.1093/annonc/mdp069. Epub 2009 Jun 23. PMID 19549707
- [Background] Homs MY, v d Gaast A, Siersema PD, Steyerberg EW, Kuipers EJ. Chemotherapy for metastatic carcinoma of the esophagus and gastro-esophageal junction. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD004063. doi: 10.1002/14651858.CD004063.pub2. PMID 17054195
- [Background] Medical Research Council Oesophageal Cancer Working Group. Surgical resection with or without preoperative chemotherapy in oesophageal cancer: a randomised controlled trial. Lancet. 2002 May 18;359(9319):1727-33. doi: 10.1016/S0140-6736(02)08651-8. PMID 12049861
- [Derived] Moehler M, Maderer A, Thuss-Patience PC, Brenner B, Meiler J, Ettrich TJ, Hofheinz RD, Al-Batran SE, Vogel A, Mueller L, Lutz MP, Lordick F, Alsina M, Borchert K, Greil R, Eisterer W, Schad A, Slotta-Huspenina J, Van Cutsem E, Lorenzen S. Cisplatin and 5-fluorouracil with or without epidermal growth factor receptor inhibition panitumumab for patients with non-resectable, advanced or metastatic oesophageal squamous cell cancer: a prospective, open-label, randomised phase III AIO/EORTC trial (POWER). Ann Oncol. 2020 Feb;31(2):228-235. doi: 10.1016/j.annonc.2019.10.018. Epub 2019 Dec 16. PMID 31959339
- See also: Related Info — http://www.aio-portal.de